CLINICAL TRIAL: NCT07135661
Title: A Prospective Phase II Randomized Controlled Trial Comparing Ultra-Hypofractionated and Moderately Hypofractionated Proton Radiotherapy Following Breast-Conserving Surgery in Early-Stage Breast Cancer（UPH-BC）
Brief Title: Ultra-Hypofractionated vs. Moderately Hypofractionated Proton Therapy for Early Breast Cancer After Lumpectomy
Acronym: UPH-BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Qing Zhang,MD, Principal Investigator, Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-BCa2024-02
Record Dates: First submitted 2025-07-10; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Proton Therapy
Keywords: Ultra-Hypofractionated Irradiation; Moderately Hypofractionated Irradiation; Breast Cancer; Proton Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate hypofractionated proton radiotherapy (Active Comparator): Whole Breast Irradiation, at 40 Gy(RBE) in 15 fractions, tumor bed SIB to 48Gy(RBE)
  Interventions: Radiation: moderate hypofractionated proton radiotherapy
- ultra-hypofractionated proton radiotherapy (Experimental): Whole breast radiotherapy, 26 Gy(RBE) in 5 fractions，tumor bed boost with 10Gy(RBE) in 2 fractions.
  Interventions: Radiation: ultra-hypofractionated proton radiotherapy

INTERVENTIONS:
Radiation: moderate hypofractionated proton radiotherapy — moderate hypofractionated proton radiotherapy: Whole Breast Irradiation, at 40 Gy(RBE) in 15 fractions, tumor bed SIB to 48Gy(RBE)
  Arms: moderate hypofractionated proton radiotherapy
Radiation: ultra-hypofractionated proton radiotherapy — Ultra-hypofractionated proton radiotherapy:Whole breast radiotherapy, 26 Gy(RBE) in 5 fractions，tumor bed boost with 10Gy(RBE) in 2 fractions.
  Arms: ultra-hypofractionated proton radiotherapy

SUMMARY:
Breast-conserving surgery (BCS) followed by whole-breast irradiation (WBI) remains the standard therapeutic approach for early-stage breast cancer. Long-term follow-up data from the FAST trial (10-year analysis) demonstrated that the 28.5 Gy/5-fraction regimen exhibited comparable adverse effects to the conventional 50 Gy/25-fraction regimen, with no statistically significant differences in photographic cosmetic assessments at 2 and 5 years post-treatment. The FAST-Forward trial demonstrated comparable 5-year ipsilateral breast tumor recurrence rates (IBTR) and incidence of radiation-related toxicities between ultra-hypofractionated whole-breast irradiation (UH-WBI; 26 Gy in 5 fractions over 1 week) and moderately hypofractionated whole-breast irradiation (MH-WBI; 40 Gy in 15 fractions over 3 weeks). Additionally, no statistically significant difference in cosmetic outcomes was observed between the two regimens at the 2-year follow-up.

Proton radiotherapy enables precise dose delivery to tumor targets while minimizing radiation exposure to surrounding normal tissues, thereby reducing treatment-related toxicities. However, current clinical protocols predominantly employ conventional fractionation for proton therapy, with a paucity of robust evidence evaluating the efficacy and safety of ultra-hypofractionated proton radiotherapy in breast cancer patients. This prospective randomized controlled trial aims to establish high-level scientific evidence for the clinical application of ultra-hypofractionated proton radiotherapy following BCS, ensuring non-inferiority in oncologic control, toxicity profiles, and cosmetic preservation compared to standard regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years
2. Pathologically (cytologically or histologically) confirmed unilateral primary invasive breast carcinoma
3. Breast conserving surgery + sentinel lymph node biopsy/axillary lymph node dissection, pathological stage pT1-2N0M0，negative margins (≥ 2 mm)
4. No distant metastasis confirmed by CT, MRI, bone scan, and PET/CT
5. No prior radiation therapy to the ipsilateral chest or breast
6. ECOG 0 ~ 2 or KPS ≥ 70

Exclusion Criteria:

1. Without pathology diagnosis
2. Positive margins or close margins (< 2mm)
3. Lymph nodes or distant metastasis
4. Bilateral breast cancer or patients with a history of contralateral breast cancer
5. Prior radiation therapy to the ipsilateral chest or breast
6. Pregnancy (confirmed by serum or urine β-HCG test) or lactation

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Cosmetic Outcomes | 2 years
  Cosmetic outcomes will be assessed at 2 years after radiotherapy. Changes in breast appearance compared to baseline will be evaluated using the Breast Cancer Treatment Outcome Scale (BCTOS), independently completed by the patient, the treating physician, and a trained research assistant at each follow-up visit. Standardized photographs of the treated breast will be taken at each assessment time point and analyzed using BCCT.core software for objective cosmetic scoring.

SECONDARY OUTCOMES:
Acute and late toxicities | 5 years
  Acute radiation-induced toxicities will be assessed from the start of radiotherapy to three months after its completion. Evaluations will be performed weekly during radiotherapy and at 1 and 3 months after treatment. Late radiation-induced toxicities will be assessed every 3 months for first 2 years, every 6 months from the 3rd to the 4th year, and annually thereafter. The toxicities will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC).
Locoregional recurrence (LRR) | 5 years
  Any first recurrence confirmed by histology or cytology within the ipsilateral breast and/or regional nodes area (including supraclavicular, infraclavicular, axillary, or internal mammary lymph nodes)
Disease-free survival (DFS) | 5 years
  The duration from the date of enrollment to the first occurrence of local recurrence, distant metastases, tumor-related death, death without prior progression, or end of follow-up.
Overall survival (OS) | 5 years
  The duration from the date of enrollment to the date of death from any cause or the last follow-up.

OTHER OUTCOMES:
Quality of Life, as measured by EORTC QLQ-BR23 questionnaire | 1 years
  To compare quality of life at 1 year after radiotherapy measured by the EORTC QLQ-BR45. Raw scores are linearly converted to a 0-100 scale with higher symptom scales reflecting increased levels of symptom burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided